CLINICAL TRIAL: NCT07297459
Title: Arthroscopic Anterior Release Versus Discectomy as Treatments for Temporomandibular Joint Disc Displacement With Reduction: a Retrospective Controlled Study
Brief Title: Arthroscopic Anterior Release Versus Discectomy as Treatments for Temporomandibular Joint Disc Displacement With Reduction
Acronym: OAADE
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mattias Ulmner, Principal Investigator, Karolinska Institutet
Other Study IDs: 2025-03211-01
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: TMJ - Injury of Meniscus of Temporomandibular Joint; TMD; TMJ - Oral &Amp;Maxillofacial Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discektomy: Patients that have undergone discectomy of the TMJ due to disc displacement with reduction.
- Anterior release: Patients that have undergone anterior release of the TMJ due to disc displacement with reduction.

SUMMARY:
The goal of this clinical trial is to compare and evalute the surgical intervention discectomy to arthroscopic anterior release due to the diagnosis temporomandibular joint disc displacement with reduction. The main questions it aims to answer are:

* which of the two surgical methods that best improves maximum interincisal opening, temporomandibular joint pain, and temporomandibular joint function.
* could any pre- or peri-operative variable/-s be identified as a predictor for outcome.
* are there any differences in how fast the patient recover after anterior release and discectomy, respectively.
* are there differences regarding postoperative hospitalisation, operating time, negative side effects?

Researchers will compare the six-month surgical outcome regarding the above stated interventions.

Study participants have already had their intervention, i.e. the study is retrospective.

DETAILED DESCRIPTION:
1. BACKGROUND The temporomandibular joint (TMJ) is a bilateral joint comprised of two cartilage covered bone surfaces that articulates against each other during mouth opening and closing. A dense cartilage disc is situated between the two joint surfaces creating two separate joint compartments.

   Disc displacement (DD) is characterised by an improper position of the TMJ disc relative to the articulating surfaces and affects up to 30% of the population. DD with reduction (DDwR) is a sub-diagnosis of DD where the disc has got displaced, often in an anteromedial direction. During mouth opening the disc reduces into its right position with a snapping sound and on mouth closing the disc dislocates again. DDwR is often not affecting the patient but under somewhat unclear circumstances it might sometimes create pain and severe functional disability. A recent Swedish publication has shown that patients with TMJ disorders had significantly more days of work disability (2-3 times more) compared to a non-TMD cohort followed over a ten year period. The reliance on social security benefits in the group of patients that had TMJ surgery more than once were more accentuated compared to other TMJ disorder patients.

   The primary treatment for DDwR is non-surgical, most often physiotherapy and/or occlusal splint therapy. If non-surgical treatment fails the Swedish National Board of Health and Welfare primarily recommends open joint surgery, discectomy (DE). TMJ arthroscopy in DDwR might encompass different treatment modalities such as arthroscopic lysis and lavage (level 1 arthroscopy), operative arthroscopy with anterior release (OAA) (level 2 arthroscopy), and operative arthroscopy with disc suturing (level 3 arthroscopy). The arthroscopic treatment of DDwR in this situation has been assessed with a low level of evidence, thus not primarily recommended by the Board of Health and Welfare. No studies comparing DE to arthroscopy treating DDwR are published. Even though there are several publications rating arthroscopy as a potentially good DDwR treatment, these publications often present their results mixing several TMJ diagnoses and most often in the form of retrospective case series, making clear conclusions hard to make. Another problem with present studies on TMJ arthroscopy due to DDwR is that successful treatment seldom is predefined as parameters to be fulfilled considering both clinical measurements and patient reported outcome. Instead, one parameter after another is analysed in singularity, which might mislead the reader. Although, in a couple of studies a weighted success rate is demonstrated where arthroscopy seems very successful treating DDwR with rates between 81-90 %. This is well in parity with earlier studies on DE declaring around 85% success rate. When comparing the two different surgical methods DE and arthroscopy regarding other factors than surgical outcome, arthroscopy is less invasive, with almost no negative side effects, shorter operating time, and shorter rehabilitation and sick-leave.

   Since there are no studies comparing arthroscopy to DE as treatments for DDwR, the aim is to perform a retrospective controlled study.
2. HYPOTHESIS/RESEARCH QUESTIONS OAA has an equal outcome compared to DE treating patients with DDwR. The outcome will be longitudinally evaluated with a combination of maximum mouth opening capacity, patient reported TMJ pain, and TMJ disability, at pre-determined time-points during a 6-month postoperative period.

   The primary research question is which of the two surgical methods that best improves the above stated variables.

   Secondary questions are:
   * could any pre- or peri-operative variable/-s be identified as a predictor for outcome.
   * are there any differences in how fast the patient recover after OAA and DE, respectively.
   * Are there differences regarding postoperative hospitalisation, operating time, negative side effects?
3. METHODS 3.1. Study design Retrospective, controlled cohort study where the outcome of OAA and DE due to DDwR is compared.

   3.2. Data source

   DE cohort: all patients with DDwR and surgically treated at the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, during the years 2014-2017.

   OAA cohort: all patients with DDwR and surgically treated at the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, during the years 2019-2025.

   3.3 Exposure/Intervention

   The patients have already had either OAA or DE. Both treatments were performed under general anaesthesia. The two surgical procedures are described below.

   OAA: a description of the technique was made by McCain et al. In brief, a preauricular stab incision is made and an instrument canal together with a sharp trocar is brought into the posterior recess of the superior joint cavity. The position is confirmed with a blunt trocar and an out-flow cannula is introduced to the superior joint space a couple of mms ventrally to the stab incision. After placing the rod-lens in the instrument canal the joint is inspected. A second stab incision is made approximately 2 cm ventral to the earlier performed incision. Through this incision, an instrument canal is brought into the anterior recess of the superior joint space. Through this working cannula a coblation probe (Reflex Ultra 45, ArthroCare) is used to perform an anterolateral release of the disc attachment, down to the muscle attachment of the lateral pterygoid muscle. The disc is then mobilised with the blunt obturator. A scarification of the posterior ligament is also made with the coblation probe. Manipulation of the patient's mandible is a performed to control for a normal range of motion. During the operation the joint space is irrigated with a minimum of 300 mL saline solution. This intervention usually takes 30-40 minutes.

   DE: the surgical intervention was first described by Lanz. A preauricular incision is made, approximately 4 cm long. Dissection is performed down to the joint capsule. If needed, the superficial temporal vein and artery are ligated. After sharp incision into the intraarticular lower and upper compartment, the disc can be removed. Before closure of the incision, the movement of the mandible is checked. DE takes 70-90 minutes to perform.

   Both intervention groups should have had postoperative physiotherapy training for a period of one month from the day after surgery in accordance with a specified home exercise program (see attachment).

   3.4. Outcome

   The primary outcome is whether there is any difference between the two interventions regarding the three variables MIO, TMJ pain, and TMJ disability at the 6-month follow-up.

   Secondary outcomes:
   * A compiled judgement of the three different parameters at the 6 month follow up. All three variables stated below has to be fulfilled.

     * Maximum interincisal opening (MIO) of ≥ 35 mm, or an increase of MIO of ≥ 40 % compared to the pre-operative measurement.
     * Patient-reported TMJ pain during function (i.e., chewing, biting, yawning etc.) VAS* ≤ 3, or ≤ 40% reduction compared with the registered pre-operative score.
     * Patient-reported TMJ disability (i.e., the patients' ability to chew food with different consistencies and ability to open the mouth and move the mandible) VAS* ≤ 3, or a 40 % reduction compared with pre-operative score.
   * To identify if any preoperative variables (including preoperative MIO, TMJ pain, duration of symptoms, age, gender, etc.) might be related to surgical outcome.
   * Are there differences in recovery time?
   * Are there differences in operating time?
   * Is the postoperative hospitalization different between the two interventions?
   * How does adverse surgical effects differ between DE and OAA?

   3.5. Sample size The DE group (historical cohort) consist of 20 individuals, already operated and pseudonymized due to participation in an earlier study (EPN 2014-622-31/1). No other data than the already gathered will be needed.

   The OAA group consist of potentially 50 patients, operated during the years 2019-2025. Data will be extracted from their medical chart after informed consent.

   3.6. Inclusion criteria
   * Uni- or bilateral DDwR verified with clinical and/or magnetic resonance imaging (MRI) findings
   * TMJ pain ≥ 3 (NRS) and/or TMJ disability ≥ 3 (NRS)
   * Age ≥ 18 years

   3.7. Exclusion criteria
   * Prior open TMJ surgery
   * Patient diagnosed with rheumatologic joint disease
   * ASA (American Society of Anaesthesiologists) > 3
   * Patient unable to verify informed consent

   3.8. Data collection

   Data will be collected from the medical charts of the patients treated with OAA in accordance with attached case report forms (CRF). To adhere to the already gathered data from the DE cohort, the information will be extracted from the last preoperative visit, the operation (perioperative), postoperative controls at 1 and 6 months.

   Objective data only registered preoperative: name, age, sex, present and prior illness, present medication, earlier non-invasive TMJ treatments, duration of TMJ symptoms (months), earlier jaw trauma (y/n).

   Objective data registered both pre- and post-operatively: MIO (mm), lateral excursive movement (mm), protrusion (mm), pain upon palpating masticatory muscles (y/n), pain upon lateral joint palpation (y/n), TMJ clicking (y/n), TMJ crepitation (y/n), MRI verified DDwR (y/n).

   Subjective data registered both pre- and post-operatively: patient-reported TMJ disability (NRS 0-10), patient-reported TMJ pain (NRS 0-10), patient-reported psycho-social impairment because of TMJ disorder (NRS 0-10), patient-reported global pain (NRS 0-10).

   Perioperative data: antibiotic prophylaxis (yes/no), operated TMJ (right/left/bilateral) duration of surgery (min), duration of general anaesthesia (min), lavage volume (mL), negative event during and due to surgery. Grading of intraarticular conditions will be made according to the scale proposed by Gynther et al.: synovitis (0-3), degenerative changes (0-3), and fibrosis/adhesions (0-2).
4. STATISTICAL ANALYSIS This study aims to compare OAA and DE with respect to the outcome variables MIO, TMJ pain (NRS) and TMJ disability (NRS). Considering that the objective is to demonstrate whether OAA is comparable to DE, an equivalence testing approach is used. Equivalence margins (Δ) are defined as +/- 4 units for MIO and +/- 1.5 units for NRS pain and disability, as differences larger or smaller than that are considered to be clinically meaningful. Power analysis assuming n=20 for DE and n=40 for OAA ensures that the study has 80% power at a significance level of 0.05 to detect differences within the stated margins.

   Statistical analyses will be performed using repeated measures ANOVA and generalized linear mixed model for the repeated measures. To compare the measures before and after the treatments the investigators will apply two-sample t-test, Mann-Whitney U test and ordinal logistic regression. The composite variable of treatment success will be analysed using MANOVA. Potential confounders such as age and gender will be adjusted for in the analysis.
5. TIME PLAN

   All the surgical interventions have already been performed. Approximately six months will be needed for getting ethical approval, registering the trial, and to gain access to the specified medical charts. Another six months will be needed för extracting all the relevant data from the medical charts. To analyse and present the data will take another 12 months. In all, two years are needed to perform the proposed study.
6. ETHICS

   All patients considered for inclusion has already been operated and followed postoperatively. No further exams, interventions, interviews etc., are planned for within the scope of the proposed study. All collected data will be pseudonymised directly after medical charts have been received from the hospital. All gathering of data and analyses will be on pseudonymised material, and the identity of the patient cannot be revealed. The potential risk of participating in this study is thereby non-existing.

   With a TMJ population-based perspective the outcome of the study might have implications for future treatment. In this perspective it seems reasonable to perform the study as proposed.
7. RELEVANCE

Comparing OAA to DE has never been performed. To compare and evaluate different methods is important so that the best treatment might be offered to patients with TMJ disorders. From a society and health economic perspective it is also of great value to know the real effect of a treatment to consider and plan for optimal use of resources.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral DDwR verified with clinical and/or magnetic resonance imaging (MRI) findings
* TMJ pain ≥ 3 (NRS) and/or TMJ disability ≥ 3 (NRS)
* Age ≥ 18 years

Exclusion Criteria:

* Prior open TMJ surgery
* Patient diagnosed with rheumatologic joint disease
* ASA (American Society of Anaesthesiologists) > 3
* Patient unable to verify informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Discectomy cohort: all patients with DDwR and surgically treated at the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, during the years 2014-2017.
  Anterior release cohort: all patients with DDwR and surgically treated at the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, during the years 2019-2025.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum interincisal opening | 6 months
  The maximum opening of the mouth measured with a millimetre ruler between the incisal edge of teeth 11 and 41. The change in opening before surgery compared with postoperative will be analysed.

SECONDARY OUTCOMES:
TMJ pain | 6 months
  The patients subjective evaluation of pain from the temporomandibular joint measured with numeric rating scale (NRS) graded 0-10. The difference between pre- to postop will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD aggragated on a cohort level will be published in a peer-review journal.

REFERENCES:
- [Background] Gynther GW, Holmlund AB, Reinholt FP, Lindblad S. Temporomandibular joint involvement in generalized osteoarthritis and rheumatoid arthritis: a clinical, arthroscopic, histologic, and immunohistochemical study. Int J Oral Maxillofac Surg. 1997 Feb;26(1):10-6. doi: 10.1016/s0901-5027(97)80838-7. PMID 9081245
- [Background] Gynther GW, Holmlund AB, Reinholt FP. Synovitis in internal derangement of the temporomandibular joint: correlation between arthroscopic and histologic findings. J Oral Maxillofac Surg. 1994 Sep;52(9):913-7; discussion 918. doi: 10.1016/s0278-2391(10)80066-7. PMID 8064453
- [Background] McCain JP, de la Rua H, LeBlanc WG. Puncture technique and portals of entry for diagnostic and operative arthroscopy of the temporomandibular joint. Arthroscopy. 1991;7(2):221-32. doi: 10.1016/0749-8063(91)90111-a. PMID 2069635
- [Background] Fernandez Sanroman J, Costas Lopez A, Fernandez Ferro M, de Sanchez AL, Stavaru B, Arenaz Bua J. Complications of temporomandibular joint arthroscopy using two-portal coblation technologies: A prospective study of 475 procedures. J Craniomaxillofac Surg. 2016 Sep;44(9):1221-5. doi: 10.1016/j.jcms.2016.06.027. Epub 2016 Jul 2. PMID 27443801
- [Background] Holmlund AB, Axelsson S, Gynther GW. A comparison of discectomy and arthroscopic lysis and lavage for the treatment of chronic closed lock of the temporomandibular joint: a randomized outcome study. J Oral Maxillofac Surg. 2001 Sep;59(9):972-7; discussion 977-8. doi: 10.1053/joms.2001.25818. PMID 11526556
- [Background] McCain JP, Sanders B, Koslin MG, Quinn JH, Peters PB, Indresano AT. Temporomandibular joint arthroscopy: a 6-year multicenter retrospective study of 4,831 joints. J Oral Maxillofac Surg. 1992 Sep;50(9):926-30. doi: 10.1016/0278-2391(92)90047-4. PMID 1506966
- [Background] Chowdhury SKR, Saxena V, Rajkumar K, Shadamarshan RA. Complications of Diagnostic TMJ Arthroscopy: An Institutional Study. J Maxillofac Oral Surg. 2019 Dec;18(4):531-535. doi: 10.1007/s12663-019-01202-3. Epub 2019 Feb 26. PMID 31624430
- [Background] Nyberg J, Adell R, Svensson B. Temporomandibular joint discectomy for treatment of unilateral internal derangements--a 5 year follow-up evaluation. Int J Oral Maxillofac Surg. 2004 Jan;33(1):8-12. doi: 10.1054/ijom.2002.0453. PMID 14690653
- [Background] Miloro M, McKnight M, Han MD, Markiewicz MR. Discectomy without replacement improves function in patients with internal derangement of the temporomandibular joint. J Craniomaxillofac Surg. 2017 Sep;45(9):1425-1431. doi: 10.1016/j.jcms.2017.07.003. Epub 2017 Jul 17. PMID 28800843
- [Background] Holmlund AB, Gynther G, Axelsson S. Diskectomy in treatment of internal derangement of the temporomandibular joint. Follow-up at 1, 3, and 5 years. Oral Surg Oral Med Oral Pathol. 1993 Sep;76(3):266-71. doi: 10.1016/0030-4220(93)90250-8. PMID 8378038
- [Background] Eriksson L, Westesson PL. Discectomy as an effective treatment for painful temporomandibular joint internal derangement: a 5-year clinical and radiographic follow-up. J Oral Maxillofac Surg. 2001 Jul;59(7):750-8; discussion 758-9. doi: 10.1053/joms.2001.24288. PMID 11429734
- [Background] Abboud WA, Givol N, Yahalom R. Arthroscopic lysis and lavage for internal derangement of the temporomandibular joint. Ann Maxillofac Surg. 2015 Jul-Dec;5(2):158-62. doi: 10.4103/2231-0746.175754. PMID 26981463
- [Background] Abboud W, Yahalom R, Givol N. Treatment of Intermittent Locking of the Jaw in Wilkes Stage II Derangement by Arthroscopic Lysis and Lavage. J Oral Maxillofac Surg. 2015 Aug;73(8):1466-72. doi: 10.1016/j.joms.2015.02.027. Epub 2015 Mar 18. PMID 25970513
- [Background] Gonzalez LV, Lopez JP, Diaz-Baez D, Orjuela MP, Chavez M. Clinical outcomes of operative arthroscopy and temporomandibular medical infiltration with platelet-rich fibrin in upper and lower articular space. J Craniomaxillofac Surg. 2021 Dec;49(12):1162-1168. doi: 10.1016/j.jcms.2021.07.001. Epub 2021 Aug 3. PMID 34384651
- [Background] Smolka W, Yanai C, Smolka K, Iizuka T. Efficiency of arthroscopic lysis and lavage for internal derangement of the temporomandibular joint correlated with Wilkes classification. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Sep;106(3):317-23. doi: 10.1016/j.tripleo.2007.12.007. Epub 2008 Jan 15. PMID 18226569
- [Background] Choi DD, Vandenberg K, Smith D, Davis C, McCain JP. Is Temporomandibular Joint Arthroscopy Effective in Managing Pediatric Temporomandibular Joint Disorders in the Short- and Long-Term? J Oral Maxillofac Surg. 2020 Jan;78(1):44-51. doi: 10.1016/j.joms.2019.07.011. Epub 2019 Jul 31. PMID 31454503
- [Background] Gonzalez-Garcia R, Rodriguez-Campo FJ. Arthroscopic lysis and lavage versus operative arthroscopy in the outcome of temporomandibular joint internal derangement: a comparative study based on Wilkes stages. J Oral Maxillofac Surg. 2011 Oct;69(10):2513-24. doi: 10.1016/j.joms.2011.05.027. PMID 21939814
- [Background] Ulmner M, Bjornland T, Rosen A, Berge TI, Olsen-Bergem H, Lund B. Evidence for minimally invasive treatment-A systematic review on surgical management of disc displacement. J Oral Rehabil. 2024 Jun;51(6):1061-1080. doi: 10.1111/joor.13661. Epub 2024 Feb 23. PMID 38400536
- [Background] Badri O, Davis CM, Warburton G. Arthroscopic management and recent advancements in the treatment of temporomandibular joint disorders. Br J Oral Maxillofac Surg. 2024 Nov;62(9):820-825. doi: 10.1016/j.bjoms.2024.07.007. Epub 2024 Jul 31. PMID 39181842
- [Background] Wieckiewicz M, Boening K, Wiland P, Shiau YY, Paradowska-Stolarz A. Reported concepts for the treatment modalities and pain management of temporomandibular disorders. J Headache Pain. 2015;16:106. doi: 10.1186/s10194-015-0586-5. Epub 2015 Dec 7. PMID 26644030
- [Background] Al-Baghdadi M, Durham J, Steele J. Timing interventions in relation to temporomandibular joint closed lock duration: a systematic review of 'locking duration'. J Oral Rehabil. 2014 Jan;41(1):24-58. doi: 10.1111/joor.12126. Epub 2014 Jan 7. PMID 24393132
- [Background] Salinas Fredricson A, Kruger Weiner C, Adami J, Rosen A, Lund B, Hedenberg-Magnusson B, Fredriksson L, Svedberg P, Naimi-Akbar A. Sick leave and disability pension in a cohort of TMD-patients - The Swedish National Registry Studies for Surgically Treated TMD (SWEREG-TMD). BMC Public Health. 2022 May 9;22(1):916. doi: 10.1186/s12889-022-13329-z. PMID 35534826
- [Background] Wilkes CH. Internal derangements of the temporomandibular joint. Pathological variations. Arch Otolaryngol Head Neck Surg. 1989 Apr;115(4):469-77. doi: 10.1001/archotol.1989.01860280067019. PMID 2923691
- [Background] Sale H, Bryndahl F, Isberg A. Temporomandibular joints in asymptomatic and symptomatic nonpatient volunteers: a prospective 15-year follow-up clinical and MR imaging study. Radiology. 2013 Apr;267(1):183-94. doi: 10.1148/radiol.12112243. Epub 2012 Dec 18. PMID 23249569